CLINICAL TRIAL: NCT00300443
Title: Safety and Efficacy Study of Bimatoprost in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-031
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension | interventions — Bimatoprost

INTERVENTIONS:
Drug: bimatoprost

SUMMARY:
The purpose of this study is to assess the safety and efficacy of bimatoprost in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of glaucoma or ocular hypertension in both eyes
* Patient requires IOP-lowering drug in both eyes

Exclusion Criteria:

* Uncontrolled medical conditions
* Ocular seasonal allergies within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Lowering intraocular pressure (IOP)

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Beach, California, United States

REFERENCES:
- [Derived] Katz LJ, Cohen JS, Batoosingh AL, Felix C, Shu V, Schiffman RM. Twelve-month, randomized, controlled trial of bimatoprost 0.01%, 0.0125%, and 0.03% in patients with glaucoma or ocular hypertension. Am J Ophthalmol. 2010 Apr;149(4):661-671.e1. doi: 10.1016/j.ajo.2009.12.003. PMID 20346780